CLINICAL TRIAL: NCT05783310
Title: Effectiveness of Psychoeducation Intervention on Reducing Negative Psychological Outcomes and Enhancing Coping of Caregivers of Children With Cancer: A Randomized Controlled Trial
Brief Title: Psychoeducation Intervention for Caregivers of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lophina Phiri, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023.040
Record Dates: First submitted 2023-03-02; First posted 2023-03-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Cancer
Keywords: Anxiety; Cancer; Caregivers; Children; Coping; Depressive symptom; Health-related quality of life; Psychoeducation intervention
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: The data collection research assistant will be blinded to the participant's allocation group to avoid the risk of assessor bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Intervention (Experimental): The intervention group will receive six sessions of a psychoeducation intervention delivered face-to-face
  Interventions: Behavioral: Psychoeducation Intervention
- Control group (No Intervention): No psychoeducation intervention will be given

INTERVENTIONS:
Behavioral: Psychoeducation Intervention — The participants in the intervention group will receive six sessions of psychoeducation intervention, lasting 60 minutes per session for six weeks. The intervention will be provided face-to-face using lectures and discussions. There will also be sharing of experience by the caregivers of children with cancer and a sharing by a caregiver of a childhood cancer survivor. The group format has been chosen to enable caregivers to offer emotional support to each other. The intervention has four components: cancer education, coping skills training, stress management techniques training, and psychological support. The intervention group will also receive the usual care.
  Arms: Psychoeducation Intervention

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of the psychoeducation intervention on anxiety, depressive symptoms, coping, and HRQoL in caregivers of children with cancer.

The study is a two-arm parallel-group single-blind, randomized controlled trial that will be conducted in two hospitals in Malawi.

DETAILED DESCRIPTION:
Aim of the study To develop and implement psychoeducation intervention that meet the need of caregivers of children with cancer in Malawi.

Objectives of the study

1. To develop a psychoeducation intervention that addresses the needs of caregivers of children with cancer in Malawian culture.
2. To evaluate the effectiveness of the PEI in reducing anxiety and depressive symptoms and enhancing coping and HRQoL among caregivers of children with cancer in Malawi.

Hypotheses of the study

1. Compared with the control group, caregivers in the intervention group will have significantly lower anxiety levels immediately after the intervention, and at 3 months post-intervention.
2. Compared with the control group, caregivers in the intervention group will have significantly fewer depressive symptoms immediately after the intervention, and at 3 months post-intervention.
3. Compared with the control group, caregivers in the intervention group will have significantly better HRQoL, immediately after the intervention, and at 3 months post-intervention.
4. Compared with the control group, caregivers in the intervention group will have significantly better coping skills immediately after the intervention, and at 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will be included if the child is within the one-year post-cancer diagnosis and on treatment, the primary carer of the child, the child is aged ≤ 15 years, caregivers are above 18 years, and caregivers must have a score of more than five on GAD-7 score. A score of 5 is the cut-off point for anxiety in this questionnaire.

Exclusion Criteria:

* Caregivers of children with other co-morbidities will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Baseline
  Anxiety will be measured using the General Anxiety Disorder questionnaire (GAD-7) GAD-7 is a 7-item scale that assesses anxiety symptoms on a 4-point scale (0=not at all to 3=nearly every day). The final score is determined by summing the scores for the seven items. Scores 5, 10, and 15 represent the cut-off points for mild, moderate, and severe anxiety, respectively.
Anxiety level | Post-intervention at six weeks
  Anxiety will be measured using the General Anxiety Disorder questionnaire (GAD-7) GAD-7 is a 7-item scale that assesses anxiety symptoms on a 4-point scale (0=not at all to 3=nearly every day). The final score is determined by summing the scores for the seven items. Scores 5, 10, and 15 represent the cut-off points for mild, moderate, and severe anxiety, respectively.
Anxiety level | Three months post-intervention
  Anxiety will be measured using the General Anxiety Disorder questionnaire (GAD-7) GAD-7 is a 7-item scale that assesses anxiety symptoms on a 4-point scale (0=not at all to 3=nearly every day). The final score is determined by summing the scores for the seven items. Scores 5, 10, and 15 represent the cut-off points for mild, moderate, and severe anxiety, respectively.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, immediately after intervention and three months follow up
  Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9).The PHQ-9 is a 9-item scale that measures depressive symptoms on a 4-point scale (0=not at all to 3=nearly every day), and the final score is obtained by summing the scores for the nine items. The scores 5, 10, 15, and 20 represent cut-off points for mild depression, moderate depression, moderately severe depression, and severe depression.
Health-related quality of life | Baseline, immediately after intervention and three months follow up
  The HRQoL will be measured using the Medical Outcomes Study (MOS) 12-item short-form health survey (SF-12) questionnaire. The SF-12 contains a subset of the SF-36 covering the eight dimensions of the HRQoL in two domains of physical health component (PHC) and mental health component (MHC). The final score is calculated by transforming each scale into 0-100; the higher the mean score, the better the HRQoL.
Coping | Baseline, immediately after intervention and three months follow up
  The coping will be measured by Brief Coping Orientation to Problems Experienced (COPE). Brief-COPE is a 28-self-reporting item scale for assessing an individual's ways of coping with stress. The tool is evaluated on the Likert scale of 1 to 4 (1 = I have not been doing it, and 4 = I have been doing it). Brief COPE has 14 subscales: active coping, use of information support, positive reframing, planning, emotional support, venting, humor, acceptance, religion, self-blame, denial, substance use, and behavioral disengagement. The total score is obtained by summing up the individual subscale; the higher score indicates high utilization of coping style in that particular subscale.

CONTACTS AND LOCATIONS:
Overall Officials: William LI, Study Chair — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (2):
- Malawi (2):
  - Queen Elizabeth Central Hospital, Blantyre
  - Kamuzu Central Hospital, Lilongwe

IPD SHARING:
Plan to Share IPD: No